CLINICAL TRIAL: NCT02758106
Title: The Instantaneous Effects of High-Frequency Chest Wall Oscillation on Patients With Acute Pneumonic Respiratory Failure Receiving Mechanical Ventilation
Brief Title: HFCWO on Pneumonic Respiratory Failure
Acronym: HFCWOonAFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Ming-Lung Chuang, Associate Professor of Internal Medicine, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CS13004
Record Dates: First submitted 2016-04-24; First posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Acute Respiratory Failure; Pneumonia
Keywords: chest wall oscillation; acute respiratory failure; airway secretion
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HFCW oscillation (Active Comparator): HFCWO was performed using a Vest Airway Clearance System Model 105 (Hill-Rom, St. Paul, Minnesota). HFCWO was applied to each subject at a frequency of 10-12 Hz and a pulse pressure setting of 1-2 selected for 15 minutes. The patients receiving HFCWO were placed in a semi-upright sitting position. Following HFCWO, suction was performed immediately via an endotracheal tube.
  Changes to the initial ventilator settings during HFCWO were recorded before and at 5, 10 and 15 minutes. The variables included peak airway pressure, positive-end expiratory pressure, respiratory rate, fraction of inspired oxygen, inspiratory time, and sensitivity settings. Following HFCWO, suction was performed immediately via an endotracheal tube.
  Interventions: Device: Vest Airway Clearance System Model 105
- placebo intervention (Placebo Comparator): the patients undergoing CCPT received cup-hand percussion with the hands positioned 3 inches from the chest, striking the chest with a waving movement while they were placed in right and left decubitus positions for 5-10 minutes each. Following CCPT, suction was performed immediately via an endotracheal tube.
  Interventions: Device: placebo intervention

INTERVENTIONS:
Device: Vest Airway Clearance System Model 105 — HFCWO for 15 minutes then sputum suction.
  Other Names: HFCW oscillation; HFCWO
  Arms: HFCW oscillation
Device: placebo intervention — CCPT for 15 minutes then sputum suction.
  Other Names: CCPT; CC physical therapy
  Arms: placebo intervention

SUMMARY:
BACKGROUND: Endotracheal intubation and prolonged immobilization of patients receiving mechanical ventilation may reduce expectoration function. High frequency chest wall oscillation (HFCWO) may ameliorate airway secretion movement; however, the vigorous oscillation may influence ventilator settings and change instantaneous cardiopulmonary responses. The aim of this study was to investigate these issues. METHODS: Seventy-three patients aged >20 years who were intubated with mechanical ventilation for pneumonic respiratory failure were recruited and randomly classified into two groups (HFCWO group, n=36; and control group who received conventional chest physical therapy (CCPT), n=37). HFCWO was applied with a fixed protocol, while CCPT was conducted using standard protocols. Both groups received sputum suction after the procedure. Changes in ventilator settings and the subjects' responses were measured at pre-set intervals and compared within groups and between groups.

DETAILED DESCRIPTION:
Pneumonia may increase bronchial secretion and decrease mucociliary function, thereby causing lung atelectasis. Patients with acute pneumonic respiratory failure receiving mechanical ventilation may therefore have a large amount of pulmonary secretions, thereby worsening bronchial hygiene, oxyhemoglobin saturation and ventilation-perfusion match. Cough function is paramount for expectoration; however, coughing is not practical for patients with endotracheal intubation and sedation. High frequency chest wall oscillation (HFCWO) may dislodge airway secretions as efficiently as conventional chest physical therapy (CCPT). However, pneumonia is not currently an indication for chest physical therapy.

HFCWO compresses and relaxes the chest wall to generate an oscillated volume from the lungs, mimicking a "mini-cough" and producing shear stress at the air-mucus interface which changes the sputum rheology, thereby improving ventilation distribution, gas mixing, and forced expired volume in one second. Most studies that have reported no significant effects have focused on mortality, hospital stay, lung function or BODE (a multidimensional 10-point scale of body mass index, severity of airflow obstruction, dyspnea rated with the modified Medical Research Council, and exercise capacity evaluated with the Six-Minute Walk Distance) score. However, these outcome measurements are not associated with the immediate effects of chest physical therapy and may be affected by other factors such as disease severity.

Using the amount of sputum as the outcome measurement of HFCWO is not strongly recommended. However, immediate cardiopulmonary changes in HFCWO have not been studied in patients receiving mechanical ventilation, although this measurement is more explicit than lung function and BODE score, as they are impractical in these patients. Changes in ventilator settings caused by HFCWO are a concern when the patients receive both treatments simultaneously. The aim of this study was to investigate the effect of HFCWO on pneumonic subjects with acute respiratory failure receiving mechanical ventilation by evaluating immediate cardiopulmonary changes and changes in the initial ventilator settings.

Methods

The investigators conducted this comparative prospective randomized controlled single-blinded study at a university hospital. Adult subjects with pneumonia complicated with acute respiratory failure requiring endotracheal intubation and mechanical ventilation were consecutively recruited from a medical intensive care unit (ICU) (20-bed capacity). Pneumonia was defined as the presence of new or progressive pulmonary infiltrates and two of the following: body temperature > 38.3C or < 36C; white blood cell count > 12,000/mL or < 4,000/mL; purulent tracheal secretions without other signs of infection requiring antimicrobial treatment. Acute respiratory failure was defined as a sudden decrease in PaO2 < 60 mm Hg (or arterial oxyhemoglobin saturation < 90%) with or without PaCO2 > 45 mm Hg.17-19 All of the patients had sufficient sputum production to require the physician to order airway secretion clearance. Disease severity was assessed by Acute Physiology and Chronic Health Evaluation (APACHE) II score. Adverse events were evaluated by the investigators and reported to the institutional review board. The exclusion criteria were pregnancy, pneumothorax, manifest hemoptysis, unstable hemodynamics, increased intracranial pressure, and those undergoing major cardiac, thoracic or abdominal surgery.

All of the eligible patients had acute pneumonic respiratory failure and received endotracheal intubation and mechanical ventilation, and all signed informed consent forms. The patients were randomly allocated to the study group (HFCWO) or the control group (CCPT), as the efficacy of bronchial hygiene for both HFCWO and CCPT is comparable4. The primary investigators were blinded to which procedure the patients received. The local institutional review board of Chung Shan Medical University Hospital approved this study (No. CS13004). The experimental research was conducted in compliance with the Helsinki Declaration.

To prevent vomiting during or after chest care, all of the subjects underwent the procedure one hour before or two hours after feeding via a nasogastric tube. Inhalation therapy was performed with an aerosolized solution of 6 mL of half saline via the ventilator before HFCWO or CCPT.

HFCWO was performed using a VestTM Airway Clearance System Model 105 (Hill-Rom, St. Paul, Minnesota) connected to a vest via two flexible tubes by trained nurses who were blinded to the purpose of the study. All of the nurses had been well trained in how to perform both HFCWO and CCPT before the study, as these procedures are routinely performed by nurses at the investigators institution. HFCWO was applied to each subject at a frequency of 10-12 Hz and a pulse pressure setting of 1-2 selected from a scale ranging from 1 to 10 (arbitrary units) for 15 minutes. The patients receiving HFCWO were placed in a semi-upright sitting position, and the patients undergoing CCPT received cup-hand percussion with the hands positioned 3 inches from the chest, striking the chest with a waving movement while they were placed in right and left decubitus positions for 5-10 minutes each1. Following HFCWO or CCPT, suction was performed immediately via an endotracheal tube.

Changes to the initial ventilator settings during HFCWO were recorded by the trained nurses by checking the ventilator panel before and at 5, 10 and 15 minutes during HFCWO. The variables included peak airway pressure (Ppeak), positive-end expiratory pressure (PEEP), respiratory rate (RR), fraction of inspired oxygen (FIO2), inspiratory time, and sensitivity settings.

Changes in the patients' cardiopulmonary responses were measured before and at 5, 10 and 15 minutes during oscillation, and at 15 minutes after sputum suction. The measurement protocol for the CCPT group was the same as for the HFCWO group, except no measurements were taken at 5 or 10 minutes during percussion because it was not possible for a single nurse to perform percussion and record measurements at the same time.

Rapid shallow breathing index (RSBI) was calculated as follows:

RSBI = breathing frequency (breaths/minute)/tidal volume (liters) (1) Oxyhemoglobin saturation was measured using a pulse oximeter (SPO2). Data were presented as mean ± standard deviation (SD) or median (interquartile range). For each outcome variable, comparisons were planned a priori. A paired t or unpaired t test was used for within-group or between-group comparisons. For non-normal data, the Mann-Whitney test was used. The chi-square test or Fisher's exact test was used to compare proportions of categorical variables between the two groups. A p value less than 0.05 was considered to be statistically significant. All statistical analyses were performed using SAS software version 9.3 (SAS Institute Inc., Cary, NC) and Microcal Origin version 4.0 (Northampton, MA, USA).

ELIGIBILITY:
Inclusion Criteria:

* acute pneumonic respiratory failure and received endotracheal intubation and mechanical ventilation,
* having sufficient sputum production to require the physician to order airway secretion clearance

Exclusion Criteria:

* pregnancy
* pneumothorax
* manifest hemoptysis
* unstable hemodynamics
* increased intracranial pressure
* those undergoing major cardiac, thoracic or abdominal surgery

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
peak airway pressure | 15 minutes
  mm Hg
mean airway pressure | 15 minutes
  mm Hg
minute ventilation | 15 minutes
  liters per minute
respiratory rate | 15 minutes
  breaths per minute
tidal volume | 15 minutes
  miniliters
rapid shallow breathing index | 15 minutes
  breaths per minute/liter
SpO2 | 15 minutes

SECONDARY OUTCOMES:
FiO2= inspired oxygen fraction | 15 minutes
respiratory rate | 15 minutes
  times per minute
airway pressure setting | 15 minutes
  mm Hg
inspiratory time | 15 minutes
  second
heart rate | 15 minutes
  beat per minute
blood pressures | 15 minutes
  mm Hg

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lung Chuang, Principal Investigator — Chung Shan Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allan JS, Garrity JM, Donahue DM. High-frequency chest-wall compression during the 48 hours following thoracic surgery. Respir Care. 2009 Mar;54(3):340-3. PMID 19245727
- [Background] Chaisson KM, Walsh S, Simmons Z, Vender RL. A clinical pilot study: high frequency chest wall oscillation airway clearance in patients with amyotrophic lateral sclerosis. Amyotroph Lateral Scler. 2006 Jun;7(2):107-11. doi: 10.1080/14660820600640570. PMID 16753975
- [Background] Clinkscale D, Spihlman K, Watts P, Rosenbluth D, Kollef MH. A randomized trial of conventional chest physical therapy versus high frequency chest wall compressions in intubated and non-intubated adults. Respir Care. 2012 Feb;57(2):221-8. doi: 10.4187/respcare.01299. Epub 2011 Jul 12. PMID 21762564
- [Background] Plioplys AV, Lewis S, Kasnicka I. Pulmonary vest therapy in pediatric long-term care. J Am Med Dir Assoc. 2002 Sep-Oct;3(5):318-21. doi: 10.1097/01.JAM.0000028225.84012.3B. PMID 12807620
- [Background] McCool FD, Rosen MJ. Nonpharmacologic airway clearance therapies: ACCP evidence-based clinical practice guidelines. Chest. 2006 Jan;129(1 Suppl):250S-259S. doi: 10.1378/chest.129.1_suppl.250S. PMID 16428718
- [Background] Whitman J, Van Beusekom R, Olson S, Worm M, Indihar F. Preliminary evaluation of high-frequency chest compression for secretion clearance in mechanically ventilated patients. Respir Care. 1993 Oct;38(10):1081-7. PMID 10145892
- [Background] Jones AP, Rowe BH. Bronchopulmonary hygiene physical therapy for chronic obstructive pulmonary disease and bronchiectasis. Cochrane Database Syst Rev. 2000;(2):CD000045. doi: 10.1002/14651858.CD000045. PMID 10796474
- [Background] Zahm JM, King M, Duvivier C, Pierrot D, Girod S, Puchelle E. Role of simulated repetitive coughing in mucus clearance. Eur Respir J. 1991 Mar;4(3):311-5. PMID 1864345
- [Background] Dosman CF, Jones RL. High-frequency chest compression: a summary of the literature. Can Respir J. 2005 Jan-Feb;12(1):37-41. doi: 10.1155/2005/525813. PMID 15776126
- [Background] Darbee JC, Kanga JF, Ohtake PJ. Physiologic evidence for high-frequency chest wall oscillation and positive expiratory pressure breathing in hospitalized subjects with cystic fibrosis. Phys Ther. 2005 Dec;85(12):1278-89. PMID 16305267
- [Background] Goktalay T, Akdemir SE, Alpaydin AO, Coskun AS, Celik P, Yorgancioglu A. Does high-frequency chest wall oscillation therapy have any impact on the infective exacerbations of chronic obstructive pulmonary disease? A randomized controlled single-blind study. Clin Rehabil. 2013 Aug;27(8):710-8. doi: 10.1177/0269215513478226. Epub 2013 Mar 15. PMID 23503735
- [Background] Park H, Park J, Woo SY, Yi YH, Kim K. Effect of high-frequency chest wall oscillation on pulmonary function after pulmonary lobectomy for non-small cell lung cancer. Crit Care Med. 2012 Sep;40(9):2583-9. doi: 10.1097/CCM.0b013e318258fd6d. PMID 22732281
- [Background] Chuang ML, Lee CY, Chen YF, Huang SF, Lin IF. Revisiting Unplanned Endotracheal Extubation and Disease Severity in Intensive Care Units. PLoS One. 2015 Oct 20;10(10):e0139864. doi: 10.1371/journal.pone.0139864. eCollection 2015. PMID 26484674
- [Background] King M, Phillips DM, Gross D, Vartian V, Chang HK, Zidulka A. Enhanced tracheal mucus clearance with high frequency chest wall compression. Am Rev Respir Dis. 1983 Sep;128(3):511-5. doi: 10.1164/arrd.1983.128.3.511. PMID 6614645
- [Background] Chatburn RL. High-frequency assisted airway clearance. Respir Care. 2007 Sep;52(9):1224-35; discussion 1235-7. PMID 17716388
- [Derived] Chuang ML, Chou YL, Lee CY, Huang SF. Instantaneous responses to high-frequency chest wall oscillation in patients with acute pneumonic respiratory failure receiving mechanical ventilation: A randomized controlled study. Medicine (Baltimore). 2017 Mar;96(9):e5912. doi: 10.1097/MD.0000000000005912. PMID 28248854